CLINICAL TRIAL: NCT05361954
Title: A Phase 1b, Dose-Escalation Study of the Safety and Preliminary Efficacy of STI-1386 Oncolytic Virus in Patients With Relapsed or Refractory Solid Tumors
Brief Title: Study to Assess the Safety and Preliminary Efficacy of STI-1386 Oncolytic Virus in Relapsed or Refractory Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OV2-RRST-101
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cancer; Cancer of Pancreas; Sarcoma; Hepatic Metastasis; Solid Tumor
Keywords: Cancer; solid tumor; hepatic metastasis
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-1386 (Experimental): A dose-escalation standard 3+3 design will be utilized and a total of 3 dosing cohorts are planned, receiving up to 4 mL of 1 x 10^6 / 1 mL, 1 x 10^7 / 1 mL, or 1 x 10^8 / 1 mL.
  Interventions: Drug: STI-1386

INTERVENTIONS:
Drug: STI-1386 — Second generation oncolytic virus
  Other Names: Seprehvec

SUMMARY:
This is a Phase 1b study to assess the safety and tolerability of STI-1386, an oncolytic virus, in subjects with relapsed and refractory solid tumors (RRSTs).

DETAILED DESCRIPTION:
This is a Phase 1b, dose-ascending study to assess the safety, tolerability and recommended phase 2 dose (RP2D) of STI-1386 in subjects with relapsed and refractory solid tumors (RRSTs). STI-1386 is a second generation oncolytic virus.

This is a two-stage study, the first stage uses a single ascending dose, followed by the multiple ascending dose stage.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed extracranial solid tumors that are relapsing or refractory including locally advanced pancreatic cancer, unresectable soft tissue sarcomas, hepatic metastases due to colorectal cancer
* At least one measurable disease per Response Evaluation Criteria in Solid Tumors v. 1.1 (RECIST 1.1) with a non-nodal lesion with longest diameter ≥ 10 mm or nodal lesions with short diameter ≥ 15 mm
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* As assessed by the investigator, ≥ 3 month life expectancy
* Adequate hematologic, liver and renal function at Screening as determined by lab criteria
* Recovered < Grade 2 from all acute toxicities from previous therapy
* Has not had prior treatment with high dose corticosteroids within the 2 weeks of screening
* Is willing and able to comply with the study schedule and other protocol requirements
* Willing to follow contraception guidelines

Exclusion Criteria:

* Have a primary brain tumor
* Use of an investigational drug or local therapy or agent within 2 weeks of first dose of study drug. Current systemic chemotherapy per investigator's discretion is allowed, but no immune checkpoint inhibitors or immune modulators
* Use of anticoagulants or anti-platelet agents unless subject can safely start/stop to allow intratumoral injections
* Use of bevacizumab (Avastin) within 28 days of the STI-1386 injection
* Diagnosis of other malignancies that have required therapy in the last year or are not in complete remission. Exceptions include non-metastatic basal cell or squamous cell carcinomas of the skin, prostate cancer or cancer in situ that does not require treatment currently or is otherwise under control
* Requiring chronic systemic immunosuppressants, including steroids > 20 mg/day
* Presence of bulky disease defined as any single mass > 5 cm in greatest dimension will trigger a discussion to determine eligibility
* New York Heart Association (NYHA) Class >3 of left ventricular ejection fraction (LVEF) < 50%
* Prolonged corrected QT interval as determined by 12-lead electrocardiogram
* Has spinal cord compression or clinically unstable brain metastases within 4 weeks of first dose of study drug
* Evidence of active herpes infection and/or chronic herpes infection requiring prophylactic antiviral medication that may not be discontinued
* Has an active or recent COVID-19 infection, must have a negative RT-PCR test and not have had symptoms within 4 weeks of day 1 of study drug administration
* Any active infection requiring systemic therapy within 72 hours of injection of STI-1386, excluding anti-viral maintenance therapy for HIV
* Moderate to severe chronic obstructive pulmonary disease or other moderate to severe chronic respiratory conditions unless under treatment and stable for the 3 months of screening
* Have active human immunodeficiency virus (HIV) infection, human T-cell leukemia virus type 1 (HTLV1) infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia
* Pregnant or lactating or up to 3 months post last dose
* Underlying medical conditions that, in the opinion of the investigator and/or medical monitor will prevent the subject from participating
* Allergy to acyclovir and related anti-HSV antiviral agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | baseline through study completion at up to approximately 29 months
  Safety as assessed by incidence of AEs by type, frequency, severity, and causality using the Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5)
Incidence of immune-related adverse events (IrAEs) | baseline through study completion at up to approximately 29 months
  Safety as assessed by incidence of IrAEs by type, frequency, severity, and causality using the Common Terminology Criteria for Adverse Events, Version 5 (CTCAEv5)

SECONDARY OUTCOMES:
Preliminary Efficacy of STI-1386 | baseline through study completion at up to approximately 29 months
  Assess the preliminary efficacy of STI-1386 using the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)
Measuring Pharmacokinetic [PK] Profile | baseline through study completion at up to approximately 29 months
  STI-1386 blood plasma concentrations will be measured
Assess immunoglobulin levels | baseline through study completion at up to approximately 29 months
  Assessment of serum immunoglobulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.